CLINICAL TRIAL: NCT03250650
Title: Transcutaneous Tibial Nerve Electrical Stimulation Combined With Transvaginal Electrical Stimulation in Overactive Bladder Syndrome Treatment: Clinical Trial
Brief Title: Physiotherapy in Overactive Bladder: Electrical Stimulation Treatment
Acronym: OAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth Alves Gonçalves Ferreira, Professor, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 63041516.7.0000.0068
Record Dates: First submitted 2017-07-13; First posted 2017-08-16 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Overactive Bladder Syndrome
Keywords: Overactive Bladder; Electric Stimulation; Physical Therapy Modalities
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Group 1: will be treated receiving Transcutaneous Tibial Electric Stimulation Group 2: will be treated receiving TTNS and Transvaginal Electric Stimulation
Who Masked: Outcomes Assessor
Masking Description: All the questionnaires (OABV-8, King´s Health, Anamnesis), Function Avaliation of Pelvic Floor Muscles, before and after treatment will be conduced by other person who is not the responsable for the research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: TTNS (Active Comparator): Intervention for Group 1: transcutaneous tibial nerve electric stimulation (TTNS), using a Device Dualpex 961(Quark medical), with 2 silicone electrode in the tibial nerve path, being one on the lower border of the medial malleolus and another one, 10cm above. Once a week for 12 weeks. The parameters used on device were, 200 microseconds for pulse time and 10Hz for Frequency, during 30 minutes.
  Interventions: Device: TTNS
- Group 2: ES + TTNS (Experimental): Intervention for Group 2: transvaginal electric stimulation plus transcutaneous tibial nerve electric stimulation (ES + TTNS), using a Device Dualpex 961(Quark medical), with transvaginal electrode, located inside the vagina. Once a week for 12 weeks. The parameters used on device were 1milisecond for pulse time and 10Hz for Frequency, during 20 minutes. After transvaginal stimulation, the tibial stimulation will be applied like described on Group 1.
  Interventions: Device: ES+TTNS

INTERVENTIONS:
Device: TTNS — Transcutaneous tibial electric stimulation
  Arms: Group 1: TTNS
Device: ES+TTNS — Transvaginal electric stimulation
  Arms: Group 2: ES + TTNS

SUMMARY:
To evaluate the efficacy of combined transvaginal electrical stimulation (ES) and transcutaneous tibial nerve electrical stimulation (TTNS) in the treatment of female overactive bladder syndrome (OAB).

DETAILED DESCRIPTION:
This is a clinical trial, blind and randomized study with 86 women with OAB or Mixed Urinary Incontinence with prevalence in the OAB symptoms, who were randomly and allocated into 2 equal groups. Group 1 underwent transcutaneous tibial nerve electrical stimulation (TTNS),for 30 minutes using 10Hz for frequency and 200µs for pulse. Group 2 received a combined of Vaginal electrical stimulation (ES) using a transvaginal probe applied ,for 20 minutes using 10Hz for frequency and 1ms for pulse and tibial nerve electrical stimulation, 30 minutes at the same parameters used in Group1. Both groups were treated once a week for 12 sessions. All patients were evaluated before and after treatment by a voiding diary, King´s Health questionnaire, avaliation of pelvic floor muscle function, overactive bladder questionnaire (OABV-8).The analyzed variables included day and night time frequency, urgency and urge incontinence.

The sample calculation was based on the difference waited between 2 groups regarding the frequency improvment.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with Overactive Bladder Syndrom no neurogenic or Mixed Incontinence Urinary with overactive bladder´s predominance symptoms more than 6 months.
* Over 18 years old.
* Normal cognitive level to understand the orientations during the treatment.

Exclusion Criteria:

* Stress Urinary Incontinence
* Drugs treatment for overactive bladder
* Pregnant women
* Neurologic diseases
* Urinary infecction
* Cystocele, rectocele and uterine prolapse
* Infectious contagious diseases
* Metal implants on the hip or lower members
* Cardiac pacemaker
* Bladder tumor
* Vaginal infecction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Decreasing the numbers of urinary frequency during day and night | 1 month
  We expect that patiens will decrease the void´s number during day (under 8), and during night, recovering theirs life´s quality.

SECONDARY OUTCOMES:
Improvement of miccional urgency and urinary urgency incontinence | 2 months
  We expect that patients will get better decreasing symptoms of urinary urgency and urinary incontinence urgency consequently.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Ferreira, PhD, Principal Investigator — University of Sao Paulo; Fernanda B Giarreta, Study Chair — University of Sao Paulo
Locations (1):
- Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
There is no plan to share participant data with other researchers.